CLINICAL TRIAL: NCT04176874
Title: Robotic-assisted Diastasis of the Rectus Abdominis Muscles Repair: Evaluation of a Minimally Invasive Surgical Procedure
Brief Title: Abdominal Diastasis Repair by Robotic Surgery
Acronym: PROMA1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190484
Record Dates: First submitted 2019-10-03; First posted 2019-11-25 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Diastasis of Muscle, Other Site
Keywords: Diastasis recti; Rectus abdominis diastasis; Robotic surgical procedure
MeSH Terms: conditions — Diastasis, Muscle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diastasis of the rectus abdominis muscles: Diastasis of the rectus abdominis muscles repair using the Intuitiv SI robot
  Interventions: Procedure: Robotic-assisted diastasis of the rectus abdominis muscles repair

INTERVENTIONS:
Procedure: Robotic-assisted diastasis of the rectus abdominis muscles repair — Diastasis of the rectus abdominis muscles repair using the Intuitiv SI robot

SUMMARY:
The objective of the study is to evaluate the feasibility of a robot-assisted minimally invasive surgical technique for the management of diastasis of the rectus abdominis. The effectiveness of this robotic surgery will be evaluated on the intermuscular distance measurement above and under umbilicus using ultrasound or CT-scan imaging.

DETAILED DESCRIPTION:
This is a bi-centric, prospective, regional research.

Patients will be included in the:

* Henri Mondor University Hospital in Créteil, in the plastic and reconstructive surgery department headed by Professor Meningaud.
* Tenon University Hospital in Paris in the plastic and reconstructive surgery department of Dr. Atlan.

As part of this research, subjects will be identified as follows:

center number (3 numeric positions) - person selection order number in the center (4 numeric positions) - initial last name - initial first name This reference is unique and will be kept for the duration of the search.

A recruitment of 50 subjects is planned. (The investigator and/or monitor) will gradually complete a form, "Pre-included Patient Register", which will include all patients (initial and date of birth) who were approached to enter the study, whether finally included or not, as well as the reasons for not including them.

Patients meeting the following criteria cannot be included:

* Patients participating or having participated in the last two months in another clinical study
* Pregnant or breastfeeding patients
* Patients not using contraception
* Patients with umbilical hernia (hernia bag)
* Patients with a history of abdominal surgery by median laparotomy
* Patients with contraindications to general anesthesia
* Any other reason that, in the investigator's opinion, could interfere with the proper conduct of the study

The trial includes: an inclusion visit, a surgical hospitalization and two follow-up visits

An initial inclusion visit,[VI], which allows you to:

* check the inclusion and non-inclusion criteria explain and give consent to the patient's research participation (which will be retrieved the day before the intervention)
* carry out the ultrasound or CT-scan for the diagnosis of diastasis.

Parameters collected during this visit

* Physical examination
* Patient's medical history relevant to the trial
* Verification of compliance with inclusion and exclusion criteria
* Ultrasound or CT-scan for the diagnosis of diastasis
* Preoperative photographic plate

The surgical procedure is performed in a single step, under general anesthesia with the assistance of the Intuitiv SI robot. The patient is placed in supine position, with his arms along his body, in the Trendelenburg position with his legs down.

An antibioprophylaxis with Amoxicillin/clavulanic acid 1g/200mg IV is administered at induction.

Preoperative marking is performed to identify the palpated medial edges of the rectus abdominis, semilunar lines and costal awnings.

Three trocars are placed: a 12mm trocar, 2 to 3 fingertips above the pubis, median for the optics, a 8mm trocar in the right iliac fossa and a 8mm trocar in the left iliac fossa. Dissection is started with the finger or foam tip scissors through the opening of the median trocar to ensure that it is in the preaponeurotic plane, in front of the anterior sheath of the large rectus abdominis muscles.

The middle trocar is set up for the robot optics and insufflation of 13 mmHg CO2. The instrument trocars are then placed (8 or 5 mm depending on the robot : 8 mm for the Intuitiv Si robot). The preaponeurotic space is dissected in front of the anterior fascia of the rectus muscles to expose the white line to the umbilicus. The umbilicus is severed, it remains vascularized by the dermal network.

Then the dissection of the preaponeurotic space is continued to the xyphoid. Lateral dissection should not go more than 3cm beyond the semi lunar lines to maintain skin vascularization, limit dead spaces and seroma formation.

The anterior aponeuroses of the great rectus muscles are plicaturized by toothed wire (type QUILL PDO) from the suspubic region to the xyphoid. The umbilicus is attached to the fascia.

A redon or Blake drain 10 is placed through one of the 8mm holes. An abdominal compression dressing is applied at the end of the procedure.

Regarding surgical management and post-operative follow-up, the following parameters will be collect:

* Duration of the intervention
* Duration of hospitalization
* Drainage time
* Weight of skin resection in case of associated excess skin fat
* Occurrence of post-operative complications: seromas, haematomas, infections, thromboembolic complications, scarring disorders

Follow-up visits will take place at 1,3 and 6 months after the intervention:

They will consist of:

* an interrogation of the patient,
* the performing of:

  * a clinical examination,
  * photographs of the face and profile of the scar
  * an abdominal ultrasound. Abdominal ultrasound was used to measure the intermuscular distance at three points (xyphoid, 3 cm above and below the umbilicus, 2 cm below the umbilicus). The average intermuscular distance was calculated from these three measurements
  * a qualitative evaluation of the scar using the VAS and POSAS scale (secondary criteria)
  * a patient satisfaction assessment using VAS scale.

The main efficacy criterion is the average intermuscular distance at 3 months post-operatively obtained by averaging ultrasound measurements at the three abdominal points defined by Beer.

The secondary efficacy criteria are:

* Duration of the procedure, duration of hospitalization, duration of post-operative drainage
* Occurrence of post-operative complications (seroma or hematoma collection, thromboembolic accident, infection, scarring disorders)
* Evaluation of the scar quality evaluated by the POSAS scale
* Overall patient satisfaction with the intervention and outcome (VAS 0 to 10)

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old or older with an indication for diastasis
* Patient who has given his or her non-opposition to participation in the research
* Patient able to understand the requirements of the trial

Exclusion Criteria:

* Patients participating or having participated in the last two months in another clinical study
* Pregnant or breastfeeding patients
* Patients not using contraception
* Patients with umbilical hernia (hernia bag)
* Patients with a history of abdominal surgery by median laparotomy
* Patients with contraindications to general anesthesia
* Any other reason that, in the investigator's opinion, could interfere with the proper conduct of the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient 18 years old or older with an indication for diastasis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
Average intermuscular distance | At 3 months post surgery
  Average intermuscular distance post-operatively obtained by averaging ultrasound measurements at the three abdominal points defined by Beer.

SECONDARY OUTCOMES:
Surgery | During the surgery
  Duration of the procedure
Hospitalization | Up to 4 days
  Duration of hospitalization
Drainage | Up to 2 days
  Duration of post-operative drainage
Complications at 1 month | At 1 month
  Occurrence of post-operative complications at 1 month
Complications at 3 months | At 3 months
  Occurrence of post-operative complications at 3 months
Complications at 6 months | At 6 months
  Occurrence of post-operative complications at 6 months
Scar quality at 1 month post surgery | at 1 months
  Evaluation of the scar quality by the POSAS scale
Scar quality at 3 months post surgery | at 3 months
  Evaluation of the scar quality by the POSAS scale
Scar quality at 6 months post surgery | at 6 months
  Evaluation of the scar quality by the POSAS scale
Patient satisfaction at 1 month post surgery | At 1 month
  Overall patient satisfaction with the intervention and outcome
Patient satisfaction at 3 months post surgery | At 3 months
  Overall patient satisfaction with the intervention and outcome
Patient satisfaction at 6 months post surgery | At 6 months
  Overall patient satisfaction with the intervention and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Barbara HERSANT, Principal Investigator — APHP
Locations (1):
- Hopital Henri Mondor, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mommers EHH, Ponten JEH, Al Omar AK, de Vries Reilingh TS, Bouvy ND, Nienhuijs SW. The general surgeon's perspective of rectus diastasis. A systematic review of treatment options. Surg Endosc. 2017 Dec;31(12):4934-4949. doi: 10.1007/s00464-017-5607-9. Epub 2017 Jun 8. PMID 28597282
- [Background] Sperstad JB, Tennfjord MK, Hilde G, Ellstrom-Engh M, Bo K. Diastasis recti abdominis during pregnancy and 12 months after childbirth: prevalence, risk factors and report of lumbopelvic pain. Br J Sports Med. 2016 Sep;50(17):1092-6. doi: 10.1136/bjsports-2016-096065. Epub 2016 Jun 20. PMID 27324871
- [Background] Akram J, Matzen SH. Rectus abdominis diastasis. J Plast Surg Hand Surg. 2014 Jun;48(3):163-9. doi: 10.3109/2000656X.2013.859145. Epub 2013 Nov 21. PMID 24256310
- [Background] Orthopoulos G, Kudsi OY. Feasibility of Robotic-Assisted Transabdominal Preperitoneal Ventral Hernia Repair. J Laparoendosc Adv Surg Tech A. 2018 Apr;28(4):434-438. doi: 10.1089/lap.2017.0595. Epub 2018 Jan 2. PMID 29293068
- [Background] Sugiyama G, Chivukula S, Chung PJ, Alfonso A. Robot-Assisted Transabdominal Preperitoneal Ventral Hernia Repair. JSLS. 2015 Oct-Dec;19(4):e2015.00092. doi: 10.4293/JSLS.2015.00092. PMID 26941547
- [Background] Nahabedian MY. Management Strategies for Diastasis Recti. Semin Plast Surg. 2018 Aug;32(3):147-154. doi: 10.1055/s-0038-1661380. Epub 2018 Jul 24. PMID 30046291
- [Background] Beer GM, Schuster A, Seifert B, Manestar M, Mihic-Probst D, Weber SA. The normal width of the linea alba in nulliparous women. Clin Anat. 2009 Sep;22(6):706-11. doi: 10.1002/ca.20836. PMID 19637295
- [Background] Bellido Luque J, Bellido Luque A, Valdivia J, Suarez Grau JM, Gomez Menchero J, Garcia Moreno J, Guadalajara Jurado J. Totally endoscopic surgery on diastasis recti associated with midline hernias. The advantages of a minimally invasive approach. Prospective cohort study. Hernia. 2015 Jun;19(3):493-501. doi: 10.1007/s10029-014-1300-2. Epub 2014 Aug 21. PMID 25142493
- [Background] Driver VR, Hanft J, Fylling CP, Beriou JM; Autologel Diabetic Foot Ulcer Study Group. A prospective, randomized, controlled trial of autologous platelet-rich plasma gel for the treatment of diabetic foot ulcers. Ostomy Wound Manage. 2006 Jun;52(6):68-70, 72, 74 passim. PMID 16799184